CLINICAL TRIAL: NCT01982968
Title: Weighing Risks and Benefits of Laparoscopic Anti-Reflux Surgery in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Treatment of IPF With Laparoscopic Anti-Reflux Surgery
Acronym: WRAP-IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00049804; 1UM1HL119089 (NIH)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Pulmonary Fibrosis; Gastroesophageal Reflux
Keywords: Idiopathic pulmonary fibrosis; IPF; Gastroesophageal reflux; GER; GERD
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Gastroesophageal Reflux | interventions — Surgical Procedures, Operative; Fundoplication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Subjects to receive standard anti-reflux treatment per clinical discretion
- Surgery (Active Comparator): Subjects will receive laparoscopic fundoplication surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Full fundoplication surgery for the treatment of abnormal GER
  Other Names: Nissen fundoplication; Laparoscopic fundoplication; Laparoscopic anti-reflux surgery
  Arms: Surgery

SUMMARY:
This study will test the hypothesis that treatment with laparoscopic anti-reflux surgery in subjects with idiopathic pulmonary fibrosis (IPF) and abnormal gastroesophageal reflux (GER) will slow the decline of forced vital capacity (FVC) over 48 weeks.

DETAILED DESCRIPTION:
This protocol proposes to test the following hypothesis: Treatment with laparoscopic anti-reflux surgery in subjects with idiopathic pulmonary fibrosis (IPF) and abnormal gastroesophageal (GER) reflux will slow the decline of forced vital capacity (FVC) over 48 weeks. This study will randomize approximately 58 subjects with IPF and abnormal acid reflux on 24-hour impedance / pH monitoring to laparoscopic anti-reflux surgery or standard care (randomization ratio 1:1). Subjects will be followed for 48 weeks or until the time of lung transplantation or death.

We aim to achieve the following: determine the impact of laparoscopic anti-reflux surgery on change in FVC over 48 weeks in patients with IPF and abnormal GER; correlate the reduction in acid and non-acid reflux events with the change in FVC over 48 weeks in patients with IPF and abnormal GER; determine the safety of laparoscopic anti-reflux surgery in patients with IPF and abnormal GER; explore the impact of laparoscopic anti-reflux surgery on key secondary endpoints over 48 weeks in patients with IPF and abnormal GER; identify molecular markers of IPF disease activity and gastroesophageal reflux in biological samples from patients with IPF and abnormal GER.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of idiopathic pulmonary fibrosis
* Abnormal GER on 24-hour pH monitoring (DeMeester score > 14.7)
* Able to provide informed consent
* Willing to undergo laparoscopic anti-reflux surgery

Exclusion Criteria:

* FVC < 50% predicted
* FEV1/FVC ratio < 0.65
* Resting room air PaO2 < 60mm Hg
* Unable to walk 50 meters on 6 minute walk test
* Acute respiratory illness in last 12 weeks
* Experimental medication for IPF in last 28 days
* Listed for lung transplantation at screening
* Unable to safely undergo surgery
* History of esophageal / bariatric / gastric surgery
* History of cancer (other than non-melanoma skin cancer) in last 3 years
* Pregnant at time of screening or enrollment
* Unable to obtain pre-authorized approval from a third party payer for surgery and related costs
* Life expectancy < 48 weeks due to another illness
* BMI > 35
* Known severe pulmonary hypertension (mean pressure > 35 mm Jg on RHC; RVSP > 50 mm Hg on ECHO)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-12; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold R Collard, MD, Principal Investigator — University of California, San Francisco; Ganesh Raghu, MD, Principal Investigator — University of Washington; Kevin J Anstrom, PhD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - University of California, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] Raghu G, Pellegrini CA, Yow E, Flaherty KR, Meyer K, Noth I, Scholand MB, Cello J, Ho LA, Pipavath S, Lee JS, Lin J, Maloney J, Martinez FJ, Morrow E, Patti MG, Rogers S, Wolters PJ, Yates R, Anstrom KJ, Collard HR. Laparoscopic anti-reflux surgery for the treatment of idiopathic pulmonary fibrosis (WRAP-IPF): a multicentre, randomised, controlled phase 2 trial. Lancet Respir Med. 2018 Sep;6(9):707-714. doi: 10.1016/S2213-2600(18)30301-1. Epub 2018 Aug 9. PMID 30100404

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Surgery
Started | 29 | 29
Completed | 21 | 27
Not Completed | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Surgery | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (7.35) | 70.6 (5.97) | 69.9 (6.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 11
  Male | 19 | 28 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity (FVC)
Description: Change in FVC (in liters) between enrollment and 48 weeks.
Time Frame: Baseline and 48 weeks
Population: Randomized patients
Measure: Mean (95% Confidence Interval); unit: liters
Groups:
- Surgery: Subjects will receive laparoscopic fundoplication surgery
  Surgery: Full fundoplication surgery for the treatment of abnormal Gastroesophageal reflux (GER)
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
liters | -0.13 [-.23 to -.02] | -0.05 [-0.15 to 0.05]

2. Secondary Outcome: Change in Score From Baseline for Acid and Non-acid Reflux Events at 48 Weeks
Description: Change in acid and non-acid reflux events from baseline to week 48. All subjects answered questions related to their reflux using a Likert scale (0 = never, 1 =occasionally, 2 = sometimes, 3 = often, 4 = always).
Time Frame: Baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
score on a scale
  Do you get heartburn? | -0.65 (1.09) | -1.04 (0.95)
  Does your stomach get bloated? | -0.40 (0.82) | -0.39 (0.99)
  Do you get bitter liquid (acid) in throat? | -0.63 (1.01) | -1.13 (0.90)
  Do you burp a lot? | -0.25 (0.72) | -0.74 (1.18)

3. Secondary Outcome: Safety of Laparoscopic Anti-reflux Surgery
Description: Overall safety of laparoscopic anti-reflux surgery in patients with IPF and abnormal GER as measured by number of participants who experienced death, serious adverse event, or other (not including serious) adverse event. See Adverse Events section for additional details.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
Participants
  All Cause Mortality | 4 | 1
  Serious Adverse Events | 8 | 5
  Other (Not Including Serious) Adverse Events | 0 | 9

4. Secondary Outcome: All-cause Mortality
Description: Impact of anti-reflux surgery on all-cause mortality from enrollment to 48 weeks
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
Participants | 4 | 1

5. Secondary Outcome: Non-elective Hospitalization
Description: Impact on non-elective hospitalizations from baseline to 48 weeks.
Time Frame: Baseline and 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
Participants | 8 | 5

6. Secondary Outcome: Acute Exacerbations
Description: Impact on acute exacerbations of IPF from baseline to week 48.
Time Frame: Baseline and 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
Participants | 4 | 1

7. Secondary Outcome: University of California San Diego (UCSD) Shortness of Breath Questionnaire (SOQB) Score
Description: Change in UCSD SOQB score from baseline to week 48. The score range is 0-120. Higher scores indicate higher breathlessness.
Time Frame: Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
score on a scale | 0.69 [-6.24 to 4.86] | 0.71 [-5.62 to 4.21]

8. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Score
Description: Change in SGRQ score from baseline to week 48. The score range is 0-100. Higher scores indicate more limitations.
Time Frame: Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
score on a scale | -3.18 [-8.35 to 1.99] | 1.04 [-3.66 to 5.74]

9. Secondary Outcome: 6-minute Walk Distance
Description: Change in 6-minute walk distance from baseline to week 48
Time Frame: Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
meters | 9.13 [-14.77 to 33.02] | 16.54 [-4.80 to 37.88]

10. Secondary Outcome: Cough Visual Analog Scale (VAS)
Description: Change in VAS from baseline to week 48. The scale range is 1-100. Lower scores indicate no cough and 100 indicates the worst cough.
Time Frame: Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Surgery
Number analyzed (Participants) | 29 | 29
score on a scale | 7.15 [-2.01 to 16.31] | 4.74 [-3.14 to 12.63]

11. Secondary Outcome: High-Resolution CT (HRCT) Fibrosis Score.
Description: Change in HRCT fibrosis score from baseline to week 48. HRCT Fibrosis score is calculated as a percentage. Higher percentage indicates more fibrosis.
Time Frame: Baseline to 48 weeks
Population: Data are not available to be reported due to inability to obtain imaging data on participants and generate a score.
Arm/Group | Control | Surgery
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Control | Surgery
All-Cause Mortality (participants affected / at risk) | 4/29 | 1/29
Serious Adverse Events (participants affected / at risk) | 8/29 | 5/29
Other Adverse Events (participants affected / at risk) | 0/29 | 9/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=29) | Surgery (N=29)
Respiratory Worsening (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
gastrointestinal haemorrhave (Gastrointestinal disorders) | 0 (0) | 1 (1)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
cholecytitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 2 (2) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=29) | Surgery (N=29)
dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (4)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT01982968/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT01982968/ICF_001.pdf